CLINICAL TRIAL: NCT00981383
Title: CAROTID: CAD Randomized Omega-3 Trial In Depression
Brief Title: Treating Depression in Coronary Artery Disease With Omega-3 Fatty Acids
Acronym: CAROTID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Toronto Rehabilitation Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAROTID-2009
Record Dates: First submitted 2009-09-10; First posted 2009-09-22 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Depression
Keywords: Fatty Acids, Omega-3
MeSH Terms: conditions — Coronary Artery Disease; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Omega-3 Fatty Acid Supplement, 1.9 g ω-3 FAs daily
  Interventions: Dietary Supplement: Omega-3 Fatty Acid Supplement
- Placebo (Placebo Comparator): Matching placebo, less than 0.12 g ω-3 FAs daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid Supplement — 3 capsules (3x1g) fish oil-derived concentrated ethyl esters, providing 1.9 g omega-3 fatty acids (1.2 g EPA and 0.6 g DHA, with 0.1 g other omega-3 fatty acids)
  Arms: Treatment
Other: Placebo — 3 capsules (3x1g) of 50/50 soybean/corn oil blend containing less than 0.12 g of omega-3 fatty acids with negligible EPA and DHA
  Arms: Placebo

SUMMARY:
Depressive disorders are common in patients with Coronary Artery Disease (CAD), occurring in up to 47% of patients. Left untreated, these symptoms not only have a strong negative impact on quality-of-life, but also increase risk of future cardiac events and death. Unfortunately, about 64% of CAD patients do not respond to current antidepressant treatments. Eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are two omega-3 (ω-3) fatty acids found in fatty fish that are important for brain function. Recent evidence showed that depressed CAD patients have lower levels of EPA and DHA than non-depressed CAD patients. This information, taken together with the known roles of ω-3 fatty acids in brain function, suggests that deficiencies may contribute to depression. However, it is unknown if increasing consumption of ω-3 fatty acids would alleviate depression and improve quality of life. While intake of adequate levels of ω-3 fatty acids is difficult to obtain through diet, concentrated supplements containing EPA and DHA that are safe, readily available, and inexpensive are now obtainable in Canada. CAROTID (CAD Randomized Omega-3 Trial In Depression) will randomize patients with CAD, with and without depressive symptoms, after 6 months of cardiac rehabilitation and usual care to receive either ω-3 fatty acid supplements or placebo daily during their final 6 months of cardiac rehabilitation. The investigators hypothesize that CAD patients randomized to receive ω-3 fatty acid supplements will show greater improvement in depressive symptoms and quality-of-life over time. The investigators will also evaluate possible improvements in other important determinants of quality of life: memory and other cognitive abilities.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) poses a serious risk to the health and well-being of the elderly. Depression is common among CAD patients and has a major negative impact on treatment outcomes and life expectancy. Late-life depression is also associated with symptoms of cognitive impairment and subsequent nonresponse to medications. Coronary artery disease and depression together can detrimentally affect autonomous seniors, resulting in increased caregiver dependence and health care resource use.

Forty-seven percent of patients with CAD have depressive disorders. About 64% of these do not respond to antidepressant treatments. Recent evidence shows that depressed CAD patients have lower levels of omega-3 fatty acids than do non-depressed CAD patients. Along with the known role of omega-3 fatty acids in brain health, this suggests that deficiencies may affect depression.

Our study, CAROTID (CAD Randomized Omega-3 Trial In Depression), is a randomized, double-blind, placebo-controlled parallel group trial in persons with CAD who are attending a cardiac rehabilitation program. Patients will receive either omega-3 fatty acids supplements or placebo daily during three months of cardiac rehab. We hypothesize that patients who receive omega-3 fatty acids will show greater improvements in depressive symptoms and quality of life. This research will determine whether there is an antidepressant effect of omega-3 fatty acids in CAD patients undergoing cardiac rehabilitation. If successful, then CAROTID will provide evidence to guide health care providers in the recommendation and use of these supplements.

ELIGIBILITY:
Inclusion Criteria:

* Language (speaks and understands English)
* Between 45-80 years old
* Stable coronary artery disease (based on no hospitalization for cardiac events for at least 7 weeks prior)
* Angiographic documentation of presence and extent of coronary artery disease (number of vessels involved, extent of stenosis, etc.)
* Written, informed consent

Exclusion Criteria:

* Significant acute medical illness (sepsis, autoimmune condition, drug overdose, uncontrolled diabetes, severely disturbed liver, kidney or lung function, anemia, hypothyroidism)
* Clinically significant cognitive impairment (Mini-Mental State Examination < 24)
* Other neurologic conditions (Parkinson's disease, Huntington's chorea, history of epilepsy, birth trauma, significant traumatic brain injury, clinical stroke, progressive supranuclear paralysis, brain tumour, subdural hematoma, multiple sclerosis)
* Canadian Cardiovascular Society Class 4 (indicating unstable angina)
* Ventricular tachycardia and/or implantable cardioverter defibrillator
* Killip class greater than II (indicates high risk of mortality in post-myocardial infarction group)
* Premorbid or concurrent psychiatric diagnoses of schizophreniform or bipolar depressive disorders, current ethanol or substance abuse or any premorbid psychiatric condition requiring hospitalization
* Current use of a concentrated omega-3 fatty acid supplement, or contraindication to soybean/corn oil
* Pregnant women
* Women who become pregnant during the course of the study will be excluded immediately.
* Women of childbearing potential must be using an approved method of birth control.
* Allergies or hypersensitivity to fish
* Pre-existing bleeding disorder
* History of electroconvulsive therapy.
* Suicidal ideation or a history of suicidal ideation/attempts (determined during SCID-I at screening/baseline visits)
* Severe depression, defined by Hamilton Depression Rating score >23
* Current or history of psychotic episode or personality disorder.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale of Depression (HAM-D) | Baseline, Week 4, Week 8, Week 12

SECONDARY OUTCOMES:
Medical Outcomes Study health survey 36-item Short Form (SF-36) | Baseline, Week 4, Week 8, Week 12
Beck Depression Inventory-II (BDI-II) | Baseline, Week 4, Week 8, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lanctôt, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Nathan Herrmann, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Toronto Rehabilitation Institute, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario

REFERENCES:
- [Result] Mazereeuw G, Herrmann N, Oh PI, Ma DW, Wang CT, Kiss A, Lanctot KL. Omega-3 Fatty Acids, Depressive Symptoms, and Cognitive Performance in Patients With Coronary Artery Disease: Analyses From a Randomized, Double-Blind, Placebo-Controlled Trial. J Clin Psychopharmacol. 2016 Oct;36(5):436-44. doi: 10.1097/JCP.0000000000000565. PMID 27529771
- [Derived] Chan P, Suridjan I, Mohammad D, Herrmann N, Mazereeuw G, Hillyer LM, Ma DWL, Oh PI, Lanctot KL. Novel Phospholipid Signature of Depressive Symptoms in Patients With Coronary Artery Disease. J Am Heart Assoc. 2018 May 5;7(10):e008278. doi: 10.1161/JAHA.117.008278. PMID 29730646
- [Derived] Mazereeuw G, Herrmann N, Xu H, Blanchard AP, Figeys D, Oh PI, Bennett SA, Lanctot KL. Platelet activating factors are associated with depressive symptoms in coronary artery disease patients: a hypothesis-generating study. Neuropsychiatr Dis Treat. 2015 Sep 4;11:2309-14. doi: 10.2147/NDT.S87111. eCollection 2015. PMID 26379437